CLINICAL TRIAL: NCT06393647
Title: Relationship Between Albumin/Creatine Ratio, B12, Folate, and Frailty Index in Patients Undergoing Gastrointestinal Malignancy Surgery
Brief Title: Relationship Between Albumin/Creatine Ratio, B12, Folate, and Frailty Index
Status: Recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AnkaraEtlikYusufOzguner007
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Frailty
Keywords: Frailty Scale; Albumin/Creatine Ratio; B12; Folate
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail group: In our study, we aim to investigate the relationship between frailty status assessed using frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) and preoperative levels of Albumin/Creatinine, B12, Folate, Ferritin, Hemogram, Sedimentation Rate, and CRP in patients undergoing gastrointestinal malignancy surgery.
  Interventions: Other: Frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36)
- Non-frail group: In our study, we aim to investigate the relationship between frailty status assessed using frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) and preoperative levels of Albumin/Creatinine, B12, Folate, Ferritin, Hemogram, Sedimentation Rate, and CRP in patients undergoing gastrointestinal malignancy surgery.
  Interventions: Other: Frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36)

INTERVENTIONS:
Other: Frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) — In our study, we aim to investigate the relationship between frailty status assessed using frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) and preoperative levels of Albumin/Creatinine, B12, Folate, Ferritin, Sedimentation Rate, and CRP in patients undergoing gastrointestinal malignancy surgery.

SUMMARY:
In the literature, the relationship between frailty and various blood tests such as beta-2 microglobulin, CRP, procalcitonin, vitamin D, IL-1, and IL-6 has been investigated (2). In our study, the investigators aim to investigate the relationship between frailty status assessed using frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) and preoperative levels of Albumin/Creatinine, B12, Folate, Ferritin, hemogram, Sedimentation Rate, and CRP in patients undergoing gastrointestinal malignancy surgery. By identifying the relationship among these parameters, the investigators believe that modifiable factors contributing to frailty in patients at risk can be addressed through appropriate interventions.

DETAILED DESCRIPTION:
Frailty is a condition associated with a decline in physiological performance. Patients are categorized as healthy, pre-frail, or frail based on physiological and functional characteristics. Frailty is known to be influenced by various lifestyle factors such as socioeconomic status, psychological factors, diet, exercise, and genetic predisposition. With aging, there is an increase in cognitive and physical dysfunction, which correlates with an increase in frailty. Along with frailty, geriatric symptoms, mortality, and other negative health outcomes also increase in the elderly population. Therefore, early detection of frailty is crucial to implementing lifestyle changes aimed at improving cognitive and physical status. Various assessment scales are used to evaluate frailty, such as the Frailty Scale Version 9, Quality of Life Scale Short Form-36, and Modified 5-item frailty index (mFI-5) In the literature, the relationship between frailty and various blood tests such as beta-2 microglobulin, CRP, procalcitonin, vitamin D, IL-1, and IL-6 has been investigated (2). In our study, the investigators aim to investigate the relationship between frailty status assessed using frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) and preoperative levels of Albumin/Creatinine, B12, Folate, Ferritin,hemogram, Sedimentation Rate, and CRP in patients undergoing gastrointestinal malignancy surgery. By identifying the relationship among these parameters, the investigators believe that modifiable factors contributing to frailty in patients at risk can be addressed through appropriate interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 65 years old.
* Patients classified under ASA (American Society of Anesthesiologists) risk groups I, II, and III.
* Patients with gastrointestinal malignancy undergoing surgery

Exclusion Criteria:

* Patients who are under 65 years old.
* Patients with an ASA score of IV or higher.
* Patients who refuse to participate in the study.
* Patients undergoing emergency surgeries will be excluded from the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In our study, we aim to investigate the relationship between frailty status assessed using frailty scale forms (Frailty Scale Version 9, Quality of Life Scale Short Form-36) and preoperative levels of Albumin/Creatine, B12, Folate, Ferritin, Sedimentation Rate, and CRP in patients undergoing gastrointestinal malignancy surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Frailty Scale Version 9 | one day before surgery
  Patients' frailty status will be assessed using the Frailty Scale Version 9.There are scores between 1 and 9 on this scale. Patients with a score of 4 or above are defined as fraile.
Quality of Life Scale Short Form-36 | one day before surgery
  SF-36 is a scale to be used to evaluate quality of life.In this scoring, scoring is between 0-100. Increasing scores are considered as positive health status.

SECONDARY OUTCOMES:
Albumin/Creatine Ratio | one day before surgery
  The ratio of albumin and creatinine to each other will be measured.
B12 levels | one day before surgery
  B12 concentration will be measured
Folate levels | one day before surgery
  Folate concentration will be measured

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Yusuf, Çankaya, Ankara
  - Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle

REFERENCES:
- [Background] Kim M, Suzuki T, Kojima N, Yoshida H, Yoshida Y, Hirano H, Won CW, Kim H. Association Between Serum beta2 -Microglobulin Levels and Prevalent and Incident Physical Frailty in Community-Dwelling Older Women. J Am Geriatr Soc. 2017 Apr;65(4):e83-e88. doi: 10.1111/jgs.14733. Epub 2017 Jan 31. PMID 28140452
- [Result] Shamliyan T, Talley KM, Ramakrishnan R, Kane RL. Association of frailty with survival: a systematic literature review. Ageing Res Rev. 2013 Mar;12(2):719-36. doi: 10.1016/j.arr.2012.03.001. Epub 2012 Mar 12. PMID 22426304